CLINICAL TRIAL: NCT02673723
Title: The Application of Docozine Combined With Sufentanil for Awake Tracheal Intubation-a Multiple Center, Randomized, Controlled，Double Blinded Clinical Trial
Brief Title: The Application of Docozine Combined With Sufentanil for Awake Tracheal Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Xinqi Cheng, Clinical Professor of Anesthesia Department, The First Affiliated Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FirstHAnhuiMU
Record Dates: First submitted 2016-01-23; First posted 2016-02-04 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Awake Tracheal Intubation
Keywords: docozine
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dezocine (Experimental): Dezocine（Dez A：0.05 mg/kg，Dez B：0.1 mg/kg and Dez C：0.15 mg/kg, diluted to 5 ml respectively) is given for 10 seconds after surface anesthesia
  Interventions: Drug: Docozine
- Controlled (Placebo Comparator): The same amount of saline is given for 10 seconds after surface anesthesia
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Docozine — dezocine（Dez A：0.05 mg/kg，Dez B：0.1 mg/kg and Dez C：0.15 mg/kg, diluted to 5 ml respectively) is given for 10 seconds after surface anesthesia
  Arms: Dezocine
Drug: Saline — The same amount of saline is given for 10 seconds after surface anesthesia
  Arms: Controlled

SUMMARY:
Mortality associated with difficult airway in anesthesia is up to 30%. So, it is urgent to find a safe and effective method for intubation. Awake tracheal intubation which is used to retain spontaneous breathing is one of the important measures to ensure the safety of the patients with difficult airway in anesthesia.

Sufentanil is used to provide good analgesia and can effectively inhibit the reaction of awake tracheal intubation, however, the outstanding problem is serious respiratory depression after intravenous sufentanil injection. Few study showed that dezocine is a kappa opioid antagonist related to mild respiratory depression and can prevents sufentanil-induced cough during general anesthesia induction.It is necessary to carry out large-scale, multi-center, randomized, controlled clinical study to determine whether dezocine prevents sufentanil-induced respiratory depression and whether dezocine combined sufentanil is a safe and effective method for awake tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent；
2. Selective surgery and general anesthesia patients；
3. Age 18-65 yrs；
4. Anesthesia Society of American (ASA) Scale I~II；

Exclusion Criteria:

1. Mallampatis Ⅲ-Ⅳ；
2. Heat rate < 50 beats/minutes；
3. II-III Atrioventricular block；
4. Use of alpha agonist or antagonist within two weeks；
5. Use of opioid within 24 hours；
6. Serious heart, liver, kidney disease and cerebrovascular disease；
7. Allergic to the trial drug and other anesthesia drug contraindication；
8. Factors existed that affect language communication；
9. Any respiratory disease；
10. Unsuccessful intubation for 3 times or drop out during intubation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Sedation assessment | anesthesia induction
  Observer's assessment of alertness/sedation(OAA/S) scale is used to assess the depth of sedation during anesthesia induction
The occurrence of cough response | anesthesia induction
  The cough scale is used to assess cough response the during anesthesia induction
The variation of blood pressure | anesthesia induction
  The variation of blood pressure（mmHg) during anesthesia induction
The variation of heart rate | anesthesia induction
  The variation of heart rate(bpm）during anesthesia induction
The variation of pulse oxygen saturation | anesthesia induction
  The variation of pulse oxygen saturation(%) during anesthesia induction

SECONDARY OUTCOMES:
The occurrence of cardiovascular events | from beginning of the anesthesia to the time the patients discharge, up to 3rd day after the surgery
  The incidence of hypertension, hypotension, tachycardia and bradycardia from beginning of the anesthesia to the time the patients discharge, up to 3rd day after the surgery is recorded
The occurrence of treatment-related adverse events | from beginning of the anesthesia to the time the patients discharge, up to 3rd day after the surgery
  The incidence of treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Er Gu, PhD,MD, Principal Investigator — First affiliated Hospital of Anhui Medical University Locations: China,
Locations (4):
- China (4):
  - Anqing Municipal Hospital, Anqing, Anhui
  - Chaohu Affiliated Hospital of Anhui Medical University, Chaohu, Anhui
  - Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The second People's Hospital of Wuhu, Wuhu, Anhui

IPD SHARING:
Plan to Share IPD: Undecided